CLINICAL TRIAL: NCT06499597
Title: Investigation of Psychometric Properties of Duke Activity Score Index in Obese Individuals Candidate for Bariatric Surgery
Brief Title: Duke Activity Score Index in Obese Individuals
Status: Recruiting | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Asst Prof, Harran University
Other Study IDs: Observ
Record Dates: First submitted 2024-07-02; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — All individuals included in the study will be included in this group and evaluations will be made.

SUMMARY:
Today, obesity is a global health problem and can lead to serious health complications. Bariatric surgery is recognized as an effective treatment option to achieve long-term weight loss and health improvement in overweight or obese individuals. However, appropriate tools are needed to assess the physical activity levels of patients before and after bariatric surgery and to guide rehabilitation processes after surgery. The Duke Activity Index (DAI) is a scale used to assess activities of daily living and was developed at Duke University Medical Center. The DAI has been widely used to determine patients' physical functioning and monitor their activity levels in various health conditions and post-surgical recovery processes. The aim of this study was to evaluate the psychometric properties of the DAI and to examine whether it is an effective tool for determining physical activity levels in patients who are candidates for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index higher than 30
* No disease that may affect functional performance
* Able to adapt to the tests to be applied

Exclusion Criteria:

* Recently hospitalized due to a condition that may make it difficult to perform the test
* Inability to perform exercise tests due to neurological or musculoskeletal disorders
* Uncontrollable medical conditions (such as lung or cardiovascular disease)
* Dysfunction of the vestibular system or eyes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients who are candidates for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Duke activity status index | Baseline (10 day before surgery), Pre-surgery (1 day before surgery)
  The Duke Activity Status Index (DASI) is an assessment tool used to evaluate the functional capacity of patients.

SECONDARY OUTCOMES:
6 minute walk test | Baseline (10 day before surgery)
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Pulmonary function test | Baseline (10 day before surgery)
  Pulmonary function tests (PFTs) allow physicians to evaluate the respiratory function of their patients in many clinical situations and when there are risk factors for lung disease, occupational exposures, and pulmonary toxicity. National guidelines for the measurements and interpretation of PFT are regularly updated, and the most recent guidelines developed by the international joint Task force from the European Respiratory Society and the American Thoracic Society (EUR/ATS) were published in 2022.
  FVC, FEV1, FEV1/FVC parameters will be evaluated. In tests, patients sit with a clip on their noses. After 3 technically appropriate tests, the best-measured values are recorded and compared against reference values. The measurements obtained are recorded as a percentage relative to their ratio to the expected reference values.FEV1 measurements are recorded as a volume in ml.
mMRC (Modified Medical Research Council) Dyspnea Scale | Baseline (10 day before surgery)
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing
Hospital Anxiety and Depression Scale (HADS) | Baseline (10 day before surgery)
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). It is worth noting that items referring to depression symptoms that describe somatic aspects of depression (e.g. insomnia and weight loss) are not included in the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No